CLINICAL TRIAL: NCT01625767
Title: Tobacco Approach Avoidance Training for Smoking Cessation in Adolescent Smokers-Study 1
Brief Title: Tobacco Approach Avoidance Training for Adolescent Smokers-1
Acronym: AAT-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Suchitra Krishnan-Sarin, Associate Professor, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1103008127-1
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Tobacco Use Disorder
Keywords: Nicotine; Smoking; Adolescent; Tobacco
MeSH Terms: conditions — Tobacco Use Disorder; Smoking

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Approach Avoidance Task experiment (Experimental): Approach Avoidance Task experiment
  Interventions: Behavioral: AAT experiment

INTERVENTIONS:
Behavioral: AAT experiment — Smokers and nonsmokers complete AAT experiment

SUMMARY:
This is a two part study. Study 1 will compare Approach Avoidance Training (AAT) responses in smokers and nonsmokers in order to confirm that adolescent smokers experience cognitive bias towards tobacco-related stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 13-18 years
* Able to read and write in English.
* Smokers: Smoking 5 or more cigarettes daily for at least 6 months; Baseline urine cotinine levels > 500 ng/ml
* Nonsmokers: Never smokers; Baseline urine cotinine levels < 50 ng/ml

Exclusion Criteria:

* Current criteria for dependence on another psychoactive substance
* Current diagnosis of psychosis, major depression or panic disorder
* Regular use of any psychoactive drugs including anxiolytics and antidepressants unless the medication has been taken consistently for 2 months, is currently being monitored by a physician, and the condition for which the medication is taken is considered to be stable
* Pregnant or lactating girls, based on self report.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
automatic approach tendencies towards smoking-related stimuli | at end of AAT at Day 1
  For all AAT comparisons, the investigators will compare median scores (to minimize influence of outliers) for cigarette approach and cigarette avoid RTs. The difference between these values gives the smoking AAT-scores, which the investigators expect to not differ from zero in the non-smokers (or to show mild avoidance), while it is expect that smokers will be faster to approach than to avoid cigarettes. ANOVA models will be used to compare scores in smokers vs. nonsmokers. Regression analyses will be used to explore the relationships between impulsivity-related measures and AAT responses.
automatic approach tendencies towards smoking-related stimuli | at end of AAT at Day 8
  For all AAT comparisons, the investigators will compare median scores (to minimize influence of outliers) for cigarette approach and cigarette avoid RTs. The difference between these values gives the smoking AAT-scores, which the investigators expect to not differ from zero in the non-smokers (or to show mild avoidance), while it is expected that smokers will be faster to approach than to avoid cigarettes. ANOVA models will be used to compare scores in smokers vs. nonsmokers. Regression analyses will be used to explore the relationships between impulsivity-related measures and AAT responses.
automatic approach tendencies towards smoking-related stimuli | at end of AAT at Day 15
  For all AAT comparisons, the investigators will compare median scores (to minimize influence of outliers) for cigarette approach and cigarette avoid RTs. The difference between these values gives the smoking AAT-scores, which the investigators expect to not differ from zero in the non-smokers (or to show mild avoidance), while it is expected that smokers will be faster to approach than to avoid cigarettes. ANOVA models will be used to compare scores in smokers vs. nonsmokers. Regression analyses will be used to explore the relationships between impulsivity-related measures and AAT responses.
automatic approach tendencies towards smoking-related stimuli | at end of AAT at Day 22
  For all AAT comparisons, the investigators will compare median scores (to minimize influence of outliers) for cigarette approach and cigarette avoid RTs. The difference between these values gives the smoking AAT-scores, which the investigators expect to not differ from zero in the non-smokers (or to show mild avoidance), while it is expected that smokers will be faster to approach than to avoid cigarettes. ANOVA models will be used to compare scores in smokers vs. nonsmokers. Regression analyses will be used to explore the relationships between impulsivity-related measures and AAT responses.
automatic approach tendencies towards smoking-related stimuli | at end of AAT at Day 29
  For all AAT comparisons, the investigators will compare median scores (to minimize influence of outliers) for cigarette approach and cigarette avoid RTs. The difference between these values gives the smoking AAT-scores, which the investigators expect to not differ from zero in the non-smokers (or to show mild avoidance), while it is expected that smokers will be faster to approach than to avoid cigarettes. ANOVA models will be used to compare scores in smokers vs. nonsmokers. Regression analyses will be used to explore the relationships between impulsivity-related measures and AAT responses.

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra Krishnan-Sarin, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University, School of Medicine, Dpeartment of Psychiatry, New Haven, Connecticut, United States

REFERENCES:
- See also: Related Info — http://try.yale.edu